CLINICAL TRIAL: NCT04625660
Title: The DETOUR2 Continued Access Clinical Trial - The Detour Endovascular Technique for Long OcclUsive Fem-pop Revascularization - Continued Access Clinical Trial
Brief Title: Detour2 Continued Access Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Endologix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLN 232
Record Dates: First submitted 2020-11-05; First posted 2020-11-12 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-03

CONDITIONS: Peripheral Artery Diseases
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Single Arm (Experimental): The PQ Bypass system is used during a minimally invasive procedure to place stent grafts in the peripheral vasculature to improve blood flow.
  Interventions: Device: PQ Bypass System

INTERVENTIONS:
Device: PQ Bypass System — Intended use from CLN232 Rev A (CLN232 is the DETOUR2 Continued Access Protocol) The PQ Bypass System is intended to improve blood flow in patients with peripheral arterial disease in symptomatic femoropopliteal lesions due to chronic total occlusions ≥ 20 cm that can include de novo, restenotic, or in-stent restenotic lesions; or total lesion lengths ≥24 cm that can include chronic total occlusions or a ≥70% lesion that includes de novo, restenotic or in-stent restenosis.

SUMMARY:
Prospective, single-arm, multi-center, clinical investigation to continue to evaluate the safety and effectiveness of the PQ Bypass System to access, deliver guidewires, and implant stent grafts for a percutaneous femoropopliteal (fem-pop) bypass.

ELIGIBILITY:
General Inclusion Criteria

1. Age > 18 and ≤ 90 years of age.
2. Willing and able to provide informed consent.
3. Subject is willing to undergo all follow-up assessments according to the specified schedule over 24 months.

   Clinical Inclusion Criteria
4. Chronic, symptomatic lower limb ischemia defined as Rutherford clinical categories 3, 4, or 5.
5. Venous Clinical Severity Score < 3.
6. Subject is a suitable candidate for angiography and endovascular intervention and, if required, is eligible for standard surgical repair.

   Angiographic Inclusion Criteria
7. Symptomatic femoropopliteal chronic total occlusions ≥ 20 cm that can include de novo, restenotic, or in-stent restenotic lesions; or Symptomatic femoropopliteal lesions ≥ 24 cm (total lesion length) that can include a chronic total occlusion or a

   * 70% lesion that includes de novo, restenotic or in-stent restenosis, by investigator visual assessment.
8. Reference vessel diameter ≥ 4.5 and ≤ 6.7 mm, by investigator visual assessment.
9. Subject has a patent popliteal artery (<50% stenosis) distal to the landing zone
10. Able to successfully access the SFA origin for entry of the crossing device.
11. At least one patent infrapopliteal vessel (<50% stenosis) with run-off to the ankle or foot.
12. A significant stenosis (≥ 50%) or occlusion of an ipsilateral, inflow artery (e.g.

aortoiliac, common femoral) must be successfully treated (use of investigational treatment prohibited) prior to treatment of the target lesion. Successful treatment is defined as no complications and less than 30% residual stenosis following intervention.

General Exclusion Criteria

1. Participating in another investigational clinical study that has not reached the study endpoint or interferes with endpoints of this study
2. Anticipated life expectancy less than 1 year or medical comorbid condition(s) that could limit the subject's ability to comply with the requirements of the trial.
3. Subject has other medical, social or psychological problems that, in the opinion of the investigator, preclude them from receiving this treatment, and the procedures and evaluations pre- and post-treatment.

   Clinical Exclusion Criteria
4. History of deep vein thrombosis the target limb.
5. Thrombophlebitis, within the previous 30 days.
6. Planned or previous major amputation of the target limb.
7. Known or suspected active infection at the time of the procedure (e.g., WIfI foot infection grade 3: Severe infection. Local infection with systemic inflammatory response syndrome [SIRS]).
8. Rutherford clinical category 0, 1, 2 or 6.
9. Has acute or chronic renal disease with GFR ≤ 30 ml/min per 1.73 m2 and/or elevated serum creatinine >2.5mg/dL (220µmol/L) or on dialysis.
10. Known hypersensitivity/allergy to the investigational devices and/or required pharmacotherapy that cannot be safely managed.
11. Morbid obesity that does not allow for safe vascular access, adequate imaging, or impacts to mobility.
12. Subject has a known coagulopathy or has bleeding diatheses, thrombocytopenia with platelet count less than 100,000/microliter or INR > 1.8.
13. Any planned vascular interventions within 14 days before and/or 30 days following the index procedure (successful inflow treatment is permitted prior to enrollment).
14. Has a known history of intracranial bleeding or aneurysm, myocardial infarction or stroke within the last 3 months.
15. Subject is pregnant or breast-feeding.

    Angiographic Exclusion Criteria
16. Stent within 3 cm of SFA ostium.
17. Previous bypass surgery on the target limb that would inhibit adequate crossing proximally and distally. (e.g. the SFA artery was ligated during the bypass surgery).
18. Subject has significant disease or obstruction (≥50%) of the inflow tract that has not been successfully treated at the time of the index procedure (success measured as

    * 30% residual stenosis, without complication)
19. Presence of aneurysm or acute thrombus in the target limb.
20. Thrombolysis of the target vessel within 72 hours prior to the index procedure, where complete resolution of the thrombus was not achieved.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2024-05-14 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
Primary Safety Endpoint at 30 Days | 30 Days
  Freedom from a major adverse event (MAE) at 30 days post-procedure defined as any occurrence of the following events: Death, Clinically-Driven Target Lesion Revascularization (CD-TLR), Major Amputation of the Treated Limb, Symptomatic Deep Vein Thrombosis (DVT), or Pulmonary Embolism, or procedure-related bleeding requiring any transfusion of packed red blood cells or surgery.
Primary Effectiveness Endpoint - Patency at 12 Months | 12 Months
  The absence of clinically-driven target lesion revascularization and absence of recurrent target lesion diameter stenosis >50% by imaging (e.g., duplex ultrasound peak systolic velocity ratio of >2.5 or invasive angiography) within the stent or immediately 1 cm above or below the treated segment. When both modalities are available, angiography takes precedence.

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - The Vascular Experts, Old Saybrook, Connecticut
  - AMITA Medical Group, Elk Grove Village, Illinois
  - Sentara Norfolk, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No